CLINICAL TRIAL: NCT00593320
Title: Stereotactic Radiosurgery (SRS) for One or Two Localized Spine Metastases
Brief Title: Stereotactic Radiosurgery (SRS) for Spine Metastases
Acronym: SRS
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Due to low accrual
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 07-0658
Record Dates: First submitted 2008-01-02; First posted 2008-01-15 (Estimated); Results first posted 2015-03-04 (Estimated); Last update posted 2015-03-04 (Estimated); Status verified 2015-02

CONDITIONS: Spinal Metastases
Keywords: SRS
MeSH Terms: interventions — Radiosurgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): Low-dose arm Single-fraction Stereotactic Radiosurgery (SRS) to 14 Gy
  Interventions: Radiation: Stereotactic Radiosurgery
- 2 (Active Comparator): High-dose arm Single-fraction Stereotactic Radiosurgery (SRS) to 18Gy
  Interventions: Radiation: Stereotactic Radiosurgery

INTERVENTIONS:
Radiation: Stereotactic Radiosurgery

SUMMARY:
This study will evaluate the most effective radiation dose. Patients will be randomized (like flipping a coin) to receive either low dose stereotactic radiotherapy (defined as "14 Gy") or high dose stereotactic radiotherapy (defined as 18 Gy).

DETAILED DESCRIPTION:
This study will evaluate the pain control and the quality of life of patients with spinal metastases using stereotactic radiotherapy. Stereotactic radiotherapy is referred to as "targeted therapy". It uses special equipment to position the patient and guide the focused beams of radiation toward the cancer and away from normal surrounding tissue. This higher dose technique may work better to kill cancer cells with fewer side effects than standard radiation therapy.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent.
* Age greater than or equal to 18 years old.
* Prior histologically-proven, non-hematogenous malignancy (Specific exclusions are multiple myeloma and lymphoma).
* Radiographic evidence of one or two non-contiguous spinal metastases amenable to SRS.
* Metastatic disease must be symptomatic (causing either pain or neurologic symptoms).
* Maximum tumor size less than or equal to 5 cm.
* Zubrod performance status of less than or equal to 3.
* Life expectancy of greater than or equal to 3 months.
* Women/Men of childbearing potential must use effective contraception.

Exclusion Criteria:

* No prior radiation delivered to the involved area
* No evidence of spinal instability requiring urgent surgical intervention.
* No evidence of spinal cord compression requiring emergent surgical or radiotherapeutic intervention.
* No plans for concomitant antineoplastic therapy (including standard fractionated RT, chemotherapy, biologic, vaccine therapy, or surgery) while on this protocol except at disease progression.Concomitant is defined as within 3 days before or after radiosurgery.
* No pregnant or lactating women.
* No active systemic infection.
* No evidence of myelopathy or cauda equina syndrome on clinical evaluation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2007-09; Primary Completion 2010-03 (Actual); Study Completion 2010-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey Bradley, M.D., Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

REFERENCES:
- See also: Alvin J. Siteman Cancer Center at Barnes-Jewish Hospital and Washington University School of Medicine — http://www.siteman.wustl.edu

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study opened to participant enrollment on 11/06/2007 and closed to participants enrollment on 03/26/2010.
Groups:
- Arm 1: Low Dose: Low-dose arm Single-fraction Stereotactic Radiosurgery (SRS) to 14 Gy
- Arm 2: High Dose: High-dose arm Single-fraction Stereotactic Radiosurgery (SRS) to 18Gy
Period: Overall Study
Arm/Group | Arm 1: Low Dose | Arm 2: High Dose
Started | 1 | 1
Completed | 1 | 1
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm 1: Low Dose | Arm 2: High Dose | Total
Number analyzed (Participants) | 1 | 1 | 2
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 1 | 1 | 2
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 1 | 2
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 1 | 1 | 2

OUTCOME MEASURES:

1. Primary Outcome: Pain Control Rate as Measured by the The Brief Pain Inventory
Description: The Brief Pain Inventory (BPI) is a 17 item patient self-rating scale assessing demographic data, use of medications, as well as sensory, and reactive components of pain.
Time Frame: 6 months after completion of treatment
Population: One patient experienced disease progression and was unable to continue to complete the required questionnaires. The second patient was removed from study due to non-compliance and did not complete the required questionnaires.
Arm/Group | Arm 1: Low Dose | Arm 2: High Dose
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Local Control Rate
Description: Local control is lack of local failure. Local failure refers to the primary treated tumor after protocol therapy and corresponds to meeting both the following two criteria: 1) Increase in tumor dimension of 20% increase in the longest diameter of the target lesion tasking as reference the smallest longest diameter since the treatment started (referred to as local enlargement). 2) The measurable tumor with criteria meeting local enlargement should be avid on PET imaging (or bone scan) with uptake of a similar intensity as the pretreatment staging PET (or bone scan), or the measurable tumor should be biopsied confirming viable carcinoma.
Time Frame: 6 months after end of treatment
Population: The first patient progressed while on treatment and the second patient was removed from study due to non-compliance.
Arm/Group | Arm 1: Low Dose | Arm 2: High Dose
Number analyzed (Participants) | 0 | 0

3. Primary Outcome: Musculoskeletal Function as Measured by the Oswestry Disability Index
Description: The Oswestry Disability Index (ODI) has 10 sections (pain intensity, personal care, lifting, walking, sitting, standing, sleeping, sex life, social life, and traveling), each of which contains 6 questions detailing the effect of pain on the ability of the patient to perform activities related to the topic of each section.
Time Frame: 6 months after completion of treatment
Population: as for outcome 1
Arm/Group | Arm 1: Low Dose | Arm 2: High Dose
Number analyzed (Participants) | 0 | 0

4. Primary Outcome: Quality of Life as Measured by the FACT-CNS Questionnaire
Description: The Functional Assessment of Cancer Therapy - Central Nervous System (FACT-CNS). The FACT-CNS consists of Physical Well-Being, Social/Family Well-Being, Emotional Well-Being, Functional Well-Being, and Additional Concerns.
  Participants can choose 0 (Not At All) up to 4 (Very Much) for each question.
Time Frame: 6 months after completion of treatment
Population: as for outcome 1
Arm/Group | Arm 1: Low Dose | Arm 2: High Dose
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Arm/Group | Arm 1: Low Dose | Arm 2: High Dose
Serious Adverse Events (participants affected / at risk) | 1/1 | 0/1
Other Adverse Events (participants affected / at risk) | 1/1 | 1/1
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm 1: Low Dose (N=1) | Arm 2: High Dose (N=1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0
Diarrhea (Gastrointestinal disorders) | 1 | 0
Hypertension (Vascular disorders) | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm 1: Low Dose (N=1) | Arm 2: High Dose (N=1)
Hypertension (Vascular disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 1
Alkaline phosphatase (Investigations) | 1 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes